CLINICAL TRIAL: NCT00043966
Title: A Randomized, Open-Label Study of 800 Mg Lopinavir/200 Mg Ritonavir QD in Combination With Tenofovir and Emtricitabine Vs. 400 Mg Lopinavir /100 Mg Ritonavir BID in Combination With Tenofovir and Emtricitabine in HIV-Infected Antiretroviral Naïve Subjects
Brief Title: Study of Lopinavir, Ritonavir, Tenofovir and Emtricitabine in HIV-Infected Antiretroviral Naïve Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M02-418
Record Dates: First submitted 2002-08-15; First posted 2002-08-19 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: treatment naive
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; Tenofovir; Emtricitabine

INTERVENTIONS:
Drug: Lopinavir/ritonavir
Drug: Tenofovir DF
Drug: Emtricitabine

SUMMARY:
The purpose of this study is to compare the safety, tolerability and antiviral activity between once-daily (QD) and twice-daily (BID) dosing of lopinavir/ritonavir and to further characterize the pharmacokinetics of once-daily dosing of lopinavir/ritonavir.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* If female, subject is not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or is of childbearing potential and practicing one of the following methods of birth control: *condoms, sponge, foams, jellies, diaphragm or intrauterine device (IUD) *contraceptives (oral or parenteral) for three months prior to study drug administration) *a vasectomized partner *total abstinence from sexual intercourse
* If female, the results of a urine pregnancy test performed at screening (urine specimen obtained no earlier than 28 days prior to study drug administration) and a urine pregnancy test performed on Study Day -1 are both negative and the subject agrees to use a barrier method of contraception throughout the study.
* Subject is not breast-feeding.
* Vital signs, physical examination and laboratory results do not exhibit evidence of acute illness.
* Subject has no significant history of cardiac, renal, neurologic, psychiatric, oncologic, endocrinologic, metabolic or hepatic disease that would adversely affect his/her participating in this study.
* Subject does not require and agrees not to take any of the following medications for the duration of the study: midazolam, triazolam, terfenadine, astemizole, cisapride, pimozide, propafenone, flecainide, certain ergot derivatives (ergotamine, dihydroergotamine, ergonovine, and methylergonovine), rifampin, lovastatin, simvastatin, and St. John's wort.
* Subject agrees not to take any medication during the study, including over-the-counter medicine, herbal medications, alcohol or recreational drugs without the knowledge and permission of the principal investigator.
* Subject has a Karnofsky Score greater than or equal to 70
* Subject has not been treated for an active AIDS-defining opportunistic infection within 30 days of screening. Subjects who are on stable maintenance therapy for an opportunistic infection may be enrolled after consultation with Abbott.
* Subject is naive to antiretroviral treatment (< 7 days ARV treatment).
* Subject has a plasma HIV RNA level of greater than 1,000 copies/mL at screening.
* Subject agrees to take all doses of the lopinavir/ritonavir from the bottles provided by the sponsor (rather than take doses from a personal "dosette" box).
* Subject has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and the subject has had the opportunity to ask questions. The informed consent must be signed before any study-specific procedures are performed.

Exclusion Criteria:

* Subject has a history of an allergic reaction or significant sensitivity to lopinavir/ritonavir, tenofovir or emtricitabine or to drugs similar to study drug.
* Subject has a recent (within the past 6 months) history of drug and/or alcohol abuse.
* Subject has a positive result on the screening tests for drugs of abuse.
* Subject has a history of substance abuse or psychiatric illness that could preclude adherence with the protocol.
* Screening laboratory analyses show any of the following abnormal laboratory results: *Hemoglobin ≤ 8.0 g/dL *Absolute neutrophil count ≤ 750 cells/µL *Platelet count ≤ 50,000 per mL *ALT or AST ≥ 3.0 x Upper Limit of Normal (ULN) *Creatinine ≥ 1.5 x Upper Limit of Normal (ULN)
* Subject has received any investigational drug within 30 days prior to study drug administration.
* For any reason, subject is considered by the investigator to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-07

PRIMARY OUTCOMES:
Proportion of subjects with plasma HIV RNA level below 50 copies/mL at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Scott Brun, M.D., Study Director — Global Project Head, Antiviral Global Project Team
Locations (52):
- United States (29):
  - Phoenix Body Positive, Phoenix, Arizona
  - Pacific Oaks Research, Beverly Hills, California
  - Orange County Center for Special Immunology, Fountain Valley, California
  - Living Hope Clinical Foundation, Long Beach, California
  - AIDS Healthcare Foundation Research Center, Los Angeles, California
  - IDS Research Initiative, Altamonte Springs, Florida
  - South Florida Clinical Research, Atlantis, Florida
  - Comprehensive Care Center, Fort Lauderdale, Florida
  - Gary J. Richmond, MD, Fort Lauderdale, Florida
  - Associates in Research, Fort Myers, Florida
  - Morris, Sklaver, Mestre & Denney, M.D., PA, Plantation, Florida
  - Health Positive, Safety Harbor, Florida
  - Infectious Disease Research Institute, Inc., Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - AIDS Research Consortium of Atlanta Inc., Atlanta, Georgia
  - Donna E. Sweet, MD, Wichita, Kansas
  - Drs. Combs and Lutz, New Orleans, Louisiana
  - St. Michael's Medical Center, Newark, New Jersey
  - Polari Medical Group, New York, New York
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Akron Infectious Disease, Inc., Akron, Ohio
  - Associates in Medical and Mental Health, P.C., Tulsa, Oklahoma
  - The Research & Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Triangle Medical, Philadelphia, Pennsylvania
  - Central Texas Clinical Research, Austin, Texas
  - Joseph C. Gathe, Jr, MD, Houston, Texas
  - Southampton Medical Group, Houston, Texas
  - Hampton Roads Medical Specialists, Hampton, Virginia
- Australia (2):
  - Ground Zero Medical Centre / AIDS Research Initiative, Darlinghurst, New South Wales
  - Holdsworth House General Practice, Darlinghurst, New South Wales
- France (6):
  - Hopital Saint Louis, Paris, Cedex 10
  - Hopital Saint Antoine, Paris, Cedex 12
  - Hopital Tenon, Paris, Cedex 20
  - CHU Kremlin Bicetre, Le Kremlin-Bicêtre
  - Hopital l'Archet, Nice
  - Hopital Bichat, Paris
- Germany (2):
  - Klinik I fur Innere Medizin der Universitat zu Koln, Cologne
  - Klinikum J.W. Goethe Universitat, Frankfurt
- Tan Tock Seng Hospital, Tan Tock Seng, Singapore
- Spain (7):
  - Hospital Germans Trias I Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Hospital 12 de Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital de Mostolesi, Madrid
- United Kingdom (5):
  - Brighton General Hospital, E. Sussex
  - Royal Free Hospital, London
  - The Caldecot Centre King's Healthcare NHS Trust, London
  - St. Stephen's Centre Chelsea & Westminster Hospital, London
  - St. Mary Hospital, London

REFERENCES:
- [Derived] Podsadecki TJ, Vrijens BC, Tousset EP, Rode RA, Hanna GJ. Decreased adherence to antiretroviral therapy observed prior to transient human immunodeficiency virus type 1 viremia. J Infect Dis. 2007 Dec 15;196(12):1773-8. doi: 10.1086/523704. PMID 18190257